CLINICAL TRIAL: NCT05702112
Title: Association of Triglyceride-glucose Index With Cardiac Hemodynamics and Cardiovascular Risk Assesment in Obese Patient.
Brief Title: Association of Triglyceride-glucose Index With Cardiac Hemodynamics
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Hany, Assistant lecturer, Assiut University
Other Study IDs: TyGI in cardiac hemodynamics
Record Dates: First submitted 2023-01-19; First posted 2023-01-27 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: TyG index; Cardiac hemodynamics
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1) To estimate the prevelance of IR in obese patients based on TYG index . 2) To screen early cardiovascular abnormalities in obese asymptomatic patients using conventional echocardiography and electrocardiogram . 3) To detect association of cardiovascular hemodynamics with TyG index . Assess cardiovascular risk in obese patients .

DETAILED DESCRIPTION:
Obesity has been a health problem of growing significance all over the world; its prevalence is increasing in both developed and developing countries . According to WHO data, 39% of the global population above 18 years of age are overweight and of these, 13% are obese. Obesity is a chronic (long-term) medical disease. Both overweight (BMI >25 kg/m2) and obesity defined as a ( Body Mass Index, or BMI, of >30 kg/m2) are associated with an increased risk of cardiovascular diseases. This is a consequence on the one hand of obesity itself and on the other hand of associated medical conditions (hypertension, diabetes, insulin resistance ,stroke ,sleep apnea, osteoarthritis, gallstones, high cholesterol, gout, and certain types of cancer ) . Obesity produces a variety of hemodynamic alterations that may cause changes in cardiac morphology which predispose to left and right ventricular dysfunction. Various neurohormonal and metabolic alterations commonly associated with obesity may contribute to these abnormalities of cardiac structure and function. Cardiovascular diseases, including heart failure (HF), atrial fibrillation (AF), and coronary artery disease (CAD), are often associated with obesity. The duration of obesity has a direct impact on the incidence of cardiovascular disease.The triglyceride-glucose (TyG) index is the logarithmized product of fasting triglycerides and fasting glucose and has been proposed as the alternative indicator of IR ( with sensitivity 96.5 % and specificity 85% ) due to its relevance to lipotoxicity and glucotoxicity compared to Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), which is expensive due to insulin measurement .TyG index has demonstrated a close relationship with cardiometabolic outcomes, namely diabetes, arterial stiffness, hypertension, cardiovascular disease (CVD), stroke and obesity-related cancers in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* The study will include obese patients over two years duration ( Jan 2023 to Jan 2024 )( age above 18 years old ; written consent will be obtained )

Exclusion Criteria:

* History of heart failure or patient known to have congenital heart disease, primary or secondary myocardial disease .

Medications associated with weight gain . Patients with previous cardiac diseases (arrhythmias - valve disease). patients who have recently used glucocorticoids or antipsychotics. Patients on statins .

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: obese patients over two years duration
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
estimate the prevelance of IR in obese patients based on TYG index . | Baseline
  The triglyceride-glucose (TyG) index is the logarithmized product of fasting triglycerides and fasting glucose and has been proposed as the alternative indicator of IR ( with sensitivity 96.5 % and specificity 85% ) due to its relevance to lipotoxicity and glucotoxicity compared to Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), which is expensive due to insulin measurement
screen early cardiovascular abnormalities in obese asymptomatic patients | Baseline
  Obesity produces a variety of hemodynamic alterations that may cause changes in cardiac morphology which predispose to left and right ventricular dysfunction. Various neurohormonal and metabolic alterations commonly associated with obesity may contribute to these abnormalities of cardiac structure and function

SECONDARY OUTCOMES:
detect association of cardiovascular hemodynamics with TyG index . | Baseline
  TyG index has demonstrated a close relationship with cardiometabolic outcomes, namely diabetes, arterial stiffness, hypertension, cardiovascular disease (CVD), stroke and obesity-related cancers in previous studies.
Assess cardiovascular risk in obese patients . | Baseline
  Cardiovascular diseases, including heart failure (HF), atrial fibrillation (AF), and coronary artery disease (CAD), are often associated with obesity. The duration of obesity has a direct impact on the incidence of cardiovascular disease.

REFERENCES:
- [Background] Zhu B, Wang J, Chen K, Yan W, Wang A, Wang W, Gao Z, Tang X, Yan L, Wan Q, Luo Z, Qin G, Chen L, Mu Y. A high triglyceride glucose index is more closely associated with hypertension than lipid or glycemic parameters in elderly individuals: a cross-sectional survey from the Reaction Study. Cardiovasc Diabetol. 2020 Jul 14;19(1):112. doi: 10.1186/s12933-020-01077-6. PMID 32664945
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Guerrero-Romero F, Simental-Mendia LE, Gonzalez-Ortiz M, Martinez-Abundis E, Ramos-Zavala MG, Hernandez-Gonzalez SO, Jacques-Camarena O, Rodriguez-Moran M. The product of triglycerides and glucose, a simple measure of insulin sensitivity. Comparison with the euglycemic-hyperinsulinemic clamp. J Clin Endocrinol Metab. 2010 Jul;95(7):3347-51. doi: 10.1210/jc.2010-0288. Epub 2010 May 19. PMID 20484475
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Zhang M, Wang B, Liu Y, Sun X, Luo X, Wang C, Li L, Zhang L, Ren Y, Zhao Y, Zhou J, Han C, Zhao J, Hu D. Cumulative increased risk of incident type 2 diabetes mellitus with increasing triglyceride glucose index in normal-weight people: The Rural Chinese Cohort Study. Cardiovasc Diabetol. 2017 Mar 1;16(1):30. doi: 10.1186/s12933-017-0514-x. PMID 28249577
- [Background] Lloyd-Jones DM, Huffman MD, Karmali KN, Sanghavi DM, Wright JS, Pelser C, Gulati M, Masoudi FA, Goff DC Jr. Estimating Longitudinal Risks and Benefits From Cardiovascular Preventive Therapies Among Medicare Patients: The Million Hearts Longitudinal ASCVD Risk Assessment Tool: A Special Report From the American Heart Association and American College of Cardiology. Circulation. 2017 Mar 28;135(13):e793-e813. doi: 10.1161/CIR.0000000000000467. Epub 2016 Nov 4. PMID 27815375
- [Background] D'Agostino RB Sr, Vasan RS, Pencina MJ, Wolf PA, Cobain M, Massaro JM, Kannel WB. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation. 2008 Feb 12;117(6):743-53. doi: 10.1161/CIRCULATIONAHA.107.699579. Epub 2008 Jan 22. PMID 18212285
- See also: Obesity — https://www.nhs.uk/conditions/obesity/
- See also: FRS risk score calculator — https://reference.medscape.com/calculator/252/framingham-risk-score-2008